CLINICAL TRIAL: NCT06242678
Title: Evaluating Spinal Cord Stimulation for Stiff Person Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00098231
Record Dates: First submitted 2024-01-24; First posted 2024-02-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-06

CONDITIONS: Stiff-Person Syndrome
MeSH Terms: conditions — Stiff-Person Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SCS trial lead (Experimental): placement of spinal cord stimulator trial leads
  Interventions: Device: SCS trial lead

INTERVENTIONS:
Device: SCS trial lead — placement of spinal cord stimulator trial leads to see if effective in the management of symptoms associated with stiff person syndrome

SUMMARY:
The purpose of this prospective pilot study is to gather preliminary evidence evaluating spinal cord stimulation (SCS) as a potential therapy for the treatment of rigidity and painful spasms in patients with stiff person syndrome (SPS), a rare autoimmune neurological condition. The hypothesis is that SCS-mediated clinical improvement occurs through multi-modal mechanisms of action targeting several components of neuronal inhibitory signaling pathways in the spinal cord.

DETAILED DESCRIPTION:
The hypothesis is that SCS-mediated clinical improvement occurs through multi-modal mechanisms of action targeting several components of neuronal inhibitory signaling pathways in the spinal cord.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years of age or older at the time that the Informed Consent Form (ICF) is signed.
* Has been clinically diagnosed with stiff person syndrome
* Has clinical symptoms of muscle rigidity and spasms in the truncal (including abdominal, thoracic paraspinal, and pectoral) or proximal lower limb musculature
* Has Cerebrospinal fluid (CSF) Anti-glutamic acid decarboxylase 65 (anti-GAD65) antibodies or serum anti-GAD65 antibodies present at any titer
* Is currently trying or has tried in the past at least two conventional therapies with insufficient symptomatic relief or intolerable side effects (such as nonsteroidal anti- inflammatory drugs, topical patches/creams/gels/ointments, physical therapy, acupuncture, bracing, assistive devices, and lifestyle modification).
* If taking oral medications, is willing to maintain a stable regimen for the duration of the study period.
* Is cleared for an implantable medical device by licensed mental health provider.
* Is an appropriate candidate for the surgical procedures required in this study based on clinical judgement of the study physician.
* Is willing to and capable of giving written informed consent.
* Is willing and able to comply with study-related requirements and procedures and attend scheduled visits.

Exclusion criteria:

* Is less than 18 years of age at the time at the time that the Informed Consent Form (ICF) is signed.
* Has a Body Mass Index (BMI) > 45.
* Has a history of spine surgery or is planning to receive a spinal injection or procedure while participating in the study, unless this procedure can be postponed until after study completion.
* Has radiological findings or evidence of moderate to severe central spinal canal stenosis or neuroforaminal stenosis at any thoracic level or laterality.
* Has radiological findings or evidence of moderate/severe central spinal canal stenosis at any cervical or lumbar level.
* Has had an epidural steroid injection within 6 weeks of enrollment.
* Has a history of infection of the spine within 6 months of enrollment.
* Has received intravenous immunoglobulin therapy within 30 days or is unwilling to maintain a stable regimen (no change in dosage or frequency) during the study period.
* Has a history of opioid misuse or current chronic opioid therapy.
* Has evidence of a coagulation abnormality or low platelet count (<120,000) indicated on Complete Blood Count test at screening, or has a history of abnormal bleeding, or if unable to pause anticoagulation therapy in accordance with accepted guidelines for a spinal cord stimulator trial.
* Has a current local infection at the anticipated surgical entry site, active systemic infection, or active malignancy.
* Has a medical condition or pain in other area(s) not intended to be treated in this study, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator (such as radicular pain, post-herpetic neuralgia, central canal stenosis of the cervical, thoracic or lumbar spine, critical limb ischemia due to peripheral vascular disease, or small vessel disease).
* Has a history of untreated major depressive disorder, or history of any mental health disorder with psychotic features, such as schizophrenia.
* Is pregnant (confirmed via pregnancy test) or plans on becoming pregnant during the study period.
* Has had, within six months of enrollment, a significant untreated addiction to dependency producing medications, alcohol or illicit drugs.
* Is concomitantly participating in another interventional clinical trial.
* Is involved in an injury claim for a study-related chronic pain that is under current litigation.
* Is a recipient of temporary Social Security Disability Insurance (SSDI) benefits due to study related chronic pain.
* Has a pending or approved worker's compensation claim for study-related chronic pain.
* Has low English language literacy interfering with the ability to complete study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Pain Scores | Baseline
  baseline pain will be measured on a 0-10 scale, with 10 being the worse level of pain, with improvement in pain level measured immediately prior to removal (kept in up to 10 days), with pain level reassessed at 14 days after trial leads removed to see if returned to baseline
Pain Scores | Day 24
  baseline pain will be measured on a 0-10 scale, with 10 being the worse level of pain, with improvement in pain level measured immediately prior to removal (kept in up to 10 days), with pain level reassessed at 14 days after trial leads removed to see if returned to baseline
Michigan Body map | baseline
  The Michigan Body Map (MBM) is a self-report measure to assess body areas of chronic pain with each area of pain marked is scored 1 point. Maximum score is 35.
Michigan Body Map | up to day 10
  The Michigan Body Map (MBM) is a self-report measure to assess body areas of chronic pain with each area of pain marked is scored 1 point. Maximum score is 35.
Penn Spasm Frequency and Severity Scale | Baseline
  The first component is a 5 point scale assessing the frequency with which spasms occur ranging from "0 = No spasms" to "4 = Spontaneous spasms occurring more than ten times per hour". The second component is a 3 point scale assessing the severity of spasms ranging from "1 = Mild" to "3 = Severe"
Penn Spasm Frequency and Severity Scale | up to day 10
  The first component is a 5 point scale assessing the frequency with which spasms occur ranging from "0 = No spasms" to "4 = Spontaneous spasms occurring more than ten times per hour". The second component is a 3 point scale assessing the severity of spasms ranging from "1 = Mild" to "3 = Severe"
Pain Disability Index | Baseline
  The Pain Disability Index (PDI) is a self-report questionnaire that measures the impact of pain on a person's life. The PDI is scored on a scale of 0 to 70, with higher scores indicating a greater degree of disability:
  0: No disability 10: Total disability
  The PDI is made up of seven items, each rated on a scale of 0 to 10:
  Family/home, Recreation, Social activity, Occupation, Sexual behavior, Self-care, and Life-support activity.
Pain Disability Index | up to Day 10
  The Pain Disability Index (PDI) is a self-report questionnaire that measures the impact of pain on a person's life. The PDI is scored on a scale of 0 to 70, with higher scores indicating a greater degree of disability:
  0: No disability 10: Total disability
  The PDI is made up of seven items, each rated on a scale of 0 to 10:
  Family/home, Recreation, Social activity, Occupation, Sexual behavior, Self-care, and Life-support activity.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction. There are seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty
Pittsburgh Sleep Quality Index (PSQI) | up to Day 10
  The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction. There are seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty
Fatigue Severity Scale (FSS) scores | baseline
  The FSS is a nine-item questionnaire that uses a seven-point Likert scale to score responses. The scale ranges from 1, which means "strongly disagree," to 7, which means "strongly agree". The minimum score is 9 and the maximum score is 63. A higher score indicates more severe fatigue.
Fatigue Severity Scale (FSS) scores | up to day 10
  The FSS is a nine-item questionnaire that uses a seven-point Likert scale to score responses. The scale ranges from 1, which means "strongly disagree," to 7, which means "strongly agree". The minimum score is 9 and the maximum score is 63. A higher score indicates more severe fatigue.
Patient Health Questionnaire-Depression | baseline
  The Patient Health Questionnaire-8 (PHQ-8) is a self-reported scale that measures depressive symptoms over the previous two weeks. The PHQ-8 is scored by adding up the scores for each of the eight items, which range from 0 to 3. The response options for each item are:
  0: Not at all
  1. Several days
  2. More than half the days
  3. Nearly every day
  The total score ranges from 0 to 24, with higher scores indicating more severe depressive symptoms. The PHQ-8's scoring categories are:
  0-4: No significant depressive symptoms 5-9: Mild symptoms 10-14: Moderate symptoms 15-19: Moderately severe symptoms 20-24: Severe symptoms A score of 10 or higher is considered major depression, and a score of 20 or higher is considered severe major depression
Patient Health Questionnaire-Depression | up to day 10
  The Patient Health Questionnaire-8 (PHQ-8) is a self-reported scale that measures depressive symptoms over the previous two weeks. The PHQ-8 is scored by adding up the scores for each of the eight items, which range from 0 to 3. The response options for each item are:
  0: Not at all
  1. Several days
  2. More than half the days
  3. Nearly every day
  The total score ranges from 0 to 24, with higher scores indicating more severe depressive symptoms. The PHQ-8's scoring categories are:
  0-4: No significant depressive symptoms 5-9: Mild symptoms 10-14: Moderate symptoms 15-19: Moderately severe symptoms 20-24: Severe symptoms A score of 10 or higher is considered major depression, and a score of 20 or higher is considered severe major depression
Generalized Anxiety Disorder | baseline
  The GAD-7 is a screening tool that measures the severity of anxiety. It's scored by assigning points to the response categories of "not at all", "several days", "more than half the days", and "nearly every day". The total score ranges from 0 to 21.
  0-4: Minimal anxiety, no intervention required 5-9: Mild anxiety, monitoring and follow-up recommended 10-14: Moderate anxiety, education about symptoms and therapy services recommended 15-21: Severe anxiety, therapy and medication recommended
Generalized Anxiety Disorder | up to day 10
  The GAD-7 is a screening tool that measures the severity of anxiety. It's scored by assigning points to the response categories of "not at all", "several days", "more than half the days", and "nearly every day". The total score ranges from 0 to 21.
  0-4: Minimal anxiety, no intervention required 5-9: Mild anxiety, monitoring and follow-up recommended 10-14: Moderate anxiety, education about symptoms and therapy services recommended 15-21: Severe anxiety, therapy and medication recommended
EuroQOL (EQ-5D-5L) | Baseline
  An index value of 1 represents the best possible health state, while an index value of <0 (variable) represents the worst possible health state.
EuroQOL (EQ-5D-5L) | up to Day 10
  An index value of 1 represents the best possible health state, while an index value of <0 (variable) represents the worst possible health state.

CONTACTS AND LOCATIONS:
Overall Officials: Janus S Patel, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
study results will be shared via publication
Supporting Information: Study Protocol
Time Frame: after study completion

DOCUMENTS (1):
  • Informed Consent Form (2026-01-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT06242678/ICF_000.pdf